CLINICAL TRIAL: NCT02039440
Title: Neutralizing Antibody Titers 6 Years After the Third Dose of Inactivated Japanese Encephalitis Vaccine and Projected Duration of Protection
Brief Title: 6-year Antibody Check After Third Vaccination Against Japanese Encephalitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Herwig Kollaritsch, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 311_FU2013; 2013-004366-34 (EudraCT Number)
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Post Other Specified Vaccination Encephalitis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): 1 blood draw
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — One-time blood draw

SUMMARY:
The purpose of this study is to determine whether there are persisting antibodies against Japanese Encephalitis 6 years after the last vaccination with IXIARO(R) and to adapt or confirm mathematical models accordingly.

DETAILED DESCRIPTION:
Japanese Encephalitis (JE) is a potentially devastating mosquito-borne viral disease. The JE virus (JEV), a Flavivirus, is endemic to many regions in Asia, and while JE is primarily a pediatric disease in the endemic regions, travelers from non-endemic regions to Asia are usually naïve to the virus and may be at risk for contracting JE at any age.

The present study aims to investigate antibody titers at approximately 6 years after the third dose of JE vaccine (JE-VC), in a cohort of participants from an earlier booster dose trial, to strengthen the statistical model of the duration of protection after the booster.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received a booster dose of JE-VC in study IC51-311
* Subjects who are willing to give written informed consent to participate in the trial

Exclusion Criteria:

* Subjects who received a further dose of any Japanese Encephalitis Vaccine since study IC51-311
* Severe immunosuppression (as result of medical conditions or medication) since study IC51-311, such as history of radiation therapy or cytostatic therapy
* simultaneous participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) for JEV neutralizing antibodies determined by PRNT | 1.5 years

SECONDARY OUTCOMES:
Seroprotection Rate (SPR) defined as rate of subjects with JEV neutralizing antibody titers ≥1:10 in a PRNT | 1.5 years

OTHER OUTCOMES:
Projected mean duration of protection after a booster dose of JE-VC | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Herwig Kollaritsch, Prof. Dr., Principal Investigator — Medizinische Universität Wien, Institut für Spezifische Prophylaxe und Tropenmedizin 1090 Wien, Kinderspitalgasse 15
Locations (1):
- Institute for Specific Prophylaxis and Tropical Medicine, Vienna, Kinderspitalgasse 15, Austria